CLINICAL TRIAL: NCT05231590
Title: A Non-Randomized, Three-Armed, Open-Label, Parallel-Group, Non-Inferiority Trial to Compare the Immunogenicity and Safety of an Adjuvanted Recombinant Spike Protein COVID-19 Vaccine (SpikoGen) in Children Aged 5 to <12 Years and 12 to <18 Years With Adults Aged 18 to 40 Years
Brief Title: Immunogenicity and Safety of the SpikoGen COVID-19 Vaccine in Children Aged 5 to <12 Years and 12 to <18 Years Compared With Adults Aged 18 to 40 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cinnagen (Industry)
Collaborators: Vaxine Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC.CIN.PT.PEDS; IRCT20150303021315N27 (Registry Identifier: Iranian Registry of Clinical Trials)
Record Dates: First submitted 2022-02-08; First posted 2022-02-09 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; Recombinant protein; Spike; Advax-SM; Advax; Vaccine; Adjuvant
MeSH Terms: conditions — COVID-19 | interventions — SARS-CoV-2 recombinant spike protein with delta inulin and CpG-ODN adjuvant vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Children Aged 5 to <12 Years (Other)
  Interventions: Biological: Low-dose SARS-CoV-2 recombinant spike protein + Advax-SM adjuvant
- Children Aged 12 to <18 Years (Other)
  Interventions: Biological: SARS-CoV-2 recombinant spike protein + Advax-SM adjuvant
- Adults Aged 18 to 40 Years (Other)
  Interventions: Biological: SARS-CoV-2 recombinant spike protein + Advax-SM adjuvant

INTERVENTIONS:
Biological: Low-dose SARS-CoV-2 recombinant spike protein + Advax-SM adjuvant — SARS-CoV-2 recombinant spike protein (12.5 µg) with Advax-SM adjuvant (7.5 mg) in two doses with a 21-day interval administered with intramuscular injections in the non-dominant arm
  Arms: Children Aged 5 to <12 Years
Biological: SARS-CoV-2 recombinant spike protein + Advax-SM adjuvant — SARS-CoV-2 recombinant spike protein (25 µg) with Advax-SM adjuvant (15 mg) in two doses with a 21-day interval administered with intramuscular injections in the non-dominant arm
  Arms: Adults Aged 18 to 40 Years; Children Aged 12 to <18 Years

SUMMARY:
This was a non-randomized, three-armed, open-label, parallel-group, non-inferiority trial designed to compare the immunogenicity and safety of the SpikoGen COVID-19 vaccine in children aged 5 to <12 years and 12 to <18 years with adults aged 18 to 40 years. Children aged 12 to <18 years and adults received 25 µg of the recombinant protein together with 15 mg of Advax-SM. Children aged 5 to <12 years received a half-dose of the adjuvanted vaccine. The injection was given in two doses with a 21-day interval in the deltoid muscle of the non-dominant arm. The vaccine immunogenicity was evaluated at 14 days after the second dose. Solicited adverse events were recorded for 7 days after each vaccination. Unsolicited adverse events were collected through one month after the second dose. Safety monitoring was continued through six months after the second dose in children aged 5 to <12 years and 12 to <18 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 5 and 40 years of age inclusive
* Willing and able to comply with all study requirements, including scheduled visits, interventions, and laboratory tests
* Healthy adults or adults in a stable medical condition, defined as not being hospitalized within 3 months prior to the screening visit
* Females must not be pregnant or breastfeeding
* Children with a body mass index equal to or greater than the 3rd percentile for age and sex as per the World Health Organization child growth standards

Exclusion Criteria:

* Subjects with signs of active SARS-CoV-2 infection at the screening visit.
* Subjects with epilepsy or a history of febrile seizures
* Subjects who receive immunosuppressive or cytotoxic medications.
* Subjects who have a history of severe allergic reactions (e.g., anaphylaxis) to the study vaccine, any components of the study interventions, or any pharmaceutical products.
* Subjects who have received any other investigational products within 30 days prior to the screening visit or intend to participate in any other clinical studies during the period of this study.
* Subjects who have been vaccinated with any vaccine or vaccine candidate against SARS-CoV-2.
* Subjects who have received any vaccines within 28 days prior to the screening visit or intend to receive any vaccines up to day 14 of the study.
* Subjects who have any known bleeding disorders or, in the investigator's opinion, have any contraindications for an intramuscular injection.
* Subjects who have received any blood, plasma, or immunoglobulin products from 90 days prior to the screening visit or intend to receive during the study period.
* Subjects with any condition that may increase the risk of participating in the study or may interfere with the evaluation of the primary endpoints of the study in the investigator's opinion.
* Subjects who have donated ≥450 mL of blood or blood products within 28 days prior to the screening visit.

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 581 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with seroconversion for SARS-CoV-2 neutralizing antibodies | 14 days after the second dose
  As measured by virus neutralization test; the primary aim of this study was to establish non-inferiority of the immunogenicity of SpikoGen COVID-19 vaccine in children aged 5 to <12 to that in adults

SECONDARY OUTCOMES:
Incidence of solicited adverse events | For 7 days after each dose
  Injection site pain, erythema, swelling, and induration, axillary swelling or tenderness ipsilateral to the side of injection, fever (oral temperature), headache, fatigue, myalgia, arthralgia, nausea, vomiting, and chills, as reported by the study participants on electronic diaries, and as defined using system organ classes and preferred terms of the Medical Dictionary for Regulatory Activities (MedDRA)
Incidence of unsolicited adverse events | Up to 1 month after the second dose
  As reported by the study participants on electronic diaries, and as defined using system organ classes and preferred terms of the Medical Dictionary for Regulatory Activities (MedDRA)
Incidence of serious adverse events (SAEs) and suspected unexpected serious adverse reaction (SUSARs) in children | Up to 6 months after the second dose
  As defined using system organ classes and preferred terms of the Medical Dictionary for Regulatory Activities (MedDRA)
Geometric mean fold rise (GMFR) for S1 binding IgG antibodies | 14 days after the second dose
  As measured by ELISA
Percentage of participants with seroconversion for S1 binding IgG antibodies | 14 days after the second dose
  As measured by ELISA
Geometric mean ratio (GMR) for S1 binding IgG antibodies | 14 days after the second dose
  As measured by ELISA
Geometric mean titer (GMT) for SARS-CoV-2 neutralizing antibodies | 14 days after the second dose
  As measured by virus neutralization test
Geometric mean fold rise (GMFR) for SARS-CoV-2 neutralizing antibodies | 14 days after the second dose
  As measured by virus neutralization test
Geometric mean ratio (GMR) for SARS-CoV-2 neutralizing antibodies | 14 days after the second dose
  As measured by virus neutralization test
Geometric mean concentration (GMC) for S1 binding IgG antibodies | 14 days after the second dose
  As measured by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Payam Tabarsi, M.D., Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Orchid Life Department, Orchid Pharmed Company, Tehran, Iran